CLINICAL TRIAL: NCT05453071
Title: The Effects of Cognitive Exercise Therapy Approach on Vascularization, Muscle Strength, Functionality, Anti-Inflammatory and Biopsycosocial Status in Individuals With Systemic Sclerosis
Brief Title: The Effect of Cognitive Exercise Therapy Approach in Individuals With Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Go 19/191
Record Dates: First submitted 2022-06-29; First posted 2022-07-12 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Systemic Sclerosis
Keywords: Systemic Sclerosis; Biopsychosocial model; BETY; Muscle strength; Functionality; Vascularization; Anti-inflammatory responses
MeSH Terms: conditions — Scleroderma, Systemic; Neovascularization, Pathologic

STUDY DESIGN:
Intervention Model Description: Evaluation parameters will be applied to the participants twice with an interval of 12 weeks. The first evaluation will be made if the individuals who come to the routine doctor's examination agree to participate in the study. According to being included in one of the two groups as those who decided to attend the BETY sessions that have been going on for 18 years and those who did not agree to attend the sessions; The individuals included in the BETY group (Group 1) will be evaluated on the day of the last exercise session after their participation in the 12-week exercise group, the individuals who do not agree to participate in the BETY sessions but agree to participate in the evaluations at 12-week intervals (Group 2) will be evaluated when they come 12 weeks apart for their routine controls. For patients with systemic sclerosis, the recommendations given routinely in our unit will be made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BETY Group (Active Comparator): Since 2004, group exercise sessions have been organized as a routine form of treatment for individuals diagnosed with rheumatism in the Department of Physiotherapy and Rehabilitation of Hacettepe University. The first evaluation will be made if the individuals who come to the routine doctor's examination agree to participate in the study. According to being included in one of the two groups as those who decided to attend the BETY sessions that have been going on for 18 years and those who did not agree to attend the sessions; The individuals included in the BETY group (Group 1) will be evaluated on the day of the last exercise session after their participation in the 12-week exercise group.
  Interventions: Other: Cognitive Exercise Therapy Approach (BETY)
- Control Group (No Intervention): Individuals (Group 2), who do not agree to participate in BETY sessions but agree to participate in evaluations with 12-week intervals, will be evaluated when they come for their routine check-ups at 12-week intervals, and recommendations given routinely.

INTERVENTIONS:
Other: Cognitive Exercise Therapy Approach (BETY) — BETY, based on function-oriented core stabilization exercises, will be applied in patients with systemic sclerosis. This exercise model includes pain management strategies, dance therapy-authentic movement. Function-oriented core stabilization exercises have the feature of being made difficult against gravity according to the person's ability to do. Initial exercises start from the stage where the distal segment of the extremity is on the ground, called closed-kinetic. This level, which is quite easy, becomes more difficult following the success of the individual. It can be started from the mat level and progressed by modifying it with theraband and exercise ball. It is used at the beginning and end of dance therapy and authentic movement sessions. In the session, cognitive restructuring technique is used to break the vicious cycle of pain-emotional-spasm during exercise. This exercise model is the main rehabilitation approach of the Rheumatological Rehabilitation Unit.
  Arms: BETY Group

SUMMARY:
The aim of this study is to investigate the effects of Cognitive Exercise Therapy Approach (BETY) on vascularization, muscle strength, functionality, anti-inflammatory and biopsychosocial status in individuals with systemic sclerosis and to present a named exercise model for this disease group with objective results.

DETAILED DESCRIPTION:
Systemic sclerosis is an inflammatory and chronic autoimmune disease. Systemic sclerosis, which was first defined by Hippocrates as thickened skin, can also progress with skin involvement and fibrosis of internal organs. Although the exact pathogenesis of the disease is not understood, it is thought to occur as a result of interactions between factors affecting collagen synthesis, fibrosis, capillary (vasculopathy) changes and immunological mechanisms. The role of inflammation has an important place in the pathogenesis of the disease. One of the most important factors governing the inflammatory process is cytokines. Changes in the response of the cytokines mentioned in systemic sclerosis, respiratory system involvement and related decrease in walking capacity, loss of muscle strength, weakening of hand functions, as well as weakening the psychological and social aspects of a person who is a biopsychosocial being. In addition to local physiotherapy applications such as paraffin applications, exercises for the face and hands, active stretching, exercise approaches such as exercises for aerobic endurance are also beneficial. However, there is no mention of a standardized exercise model, the quality of life of individuals with systemic sclerosis, which is a rare disease, activities of daily living, studies in which the social and psychological aspects of the individual are included in the treatment, and named and defined exercise methods are lacking in the literature. It is seen that studies are generally carried out with scales and functional tests.

Cognitive Exercise Therapy Approach, presents an example of an innovative biopsychosocial model with its own biopsychosocial scale, the basic exercise model of which is core stabilization exercises, including pain management, mood management and sexual information management. For individuals with systemic sclerosis, which is in the group of rare diseases, it is necessary to present the results of the intervention with objective evaluation methods to the literature. In this study, it is aimed to present an exercise model named for this disease group with objective results by examining the effects of Cognitive Exercise Therapy Approach (BETY) on vascularization, muscle strength, functionality, anti-inflammatory and biopsychosocial status in individuals with systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Systemic Sclerosis
* Being between the ages of 18-65
* Regular attendance at the rheumatology outpatient clinic at Hacettepe University
* No medication change in the last 3 months

Exclusion Criteria:

* Having a severe musculoskeletal disability Being diagnosed with pulmonary hypertension
* FVC value below 50%
* History of active infection
* Symptomatic cardiac involvement
* Having a psychiatric disorder
* Pregnancy
* History of active myositis
* Renal failure
* Not being literate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire (BETY-BQ) | 3 Months
  It is a 5-point Likert-type scale consisting of 30 questions developed with individuals with rheumatism. It is a practical scale that evaluates individuals in terms of fatigue and functionality, sleep, mood, sexuality, pain and sociability. Each question is scored as "0= never, 1=yes rarely, 2=yes sometimes, 3=yes often 4=yes always" and gives a total score over 30 items. A high score means a low biopsychosocial level. The total score is scored between 0-120

SECONDARY OUTCOMES:
Modified Rodnan Skin Score (mRSS) | 3 Months
  A method in which the skin firmness of the person is evaluated by holding the skin between two fingers and looking at the degree of stretching. It is a standard disease activity scoring applied in doctor's examinations for Systemic Sclerosis patients. It evaluates the skin hardness of 17 different parts of the body. 0= normal skin , 1= mild skin thickness, 2= moderate skin thickness, 3= severe skin thickness. A high score indicates increased skin thickness. The total score is scored between 0-51
Quality of Life Scale Short Form-36 (SF-36) | 3 Months
  SF-36 Quality of Life Scale; It is a 36-item, 11-question scale that allows general health screening with 8 sub-parameters consisting of general health, physical function, social function, pain, emotional well-being, role limitations due to physical health, role limitations due to emotional problems and vitality. It is a generic scale, Items are scored as '0 = worst health condition 100 = best health state'. Each subcategory is scored between 0 and 100 points, with a high score indicating good health.
Scleroderma Health Assessment Questionnaire (SHAQ) | 3 Months
  Dressing and grooming, arising, eating, walking, hygiene, reach, grip and activities are evaluated with 20 items divided into eight areas. The answers given to each question range from "without any difficulty (0)", "with some difficulty (1)", "with much difficulty (2)" and "unable to do (3)". Afterwards, it is requested to show how Raynaud's phenomenon, digital ulcers, intestinal involvement, respiratory and overall disease severity affect the daily activity level on a 15 cm long section. The SHAQ-global score is formed by dividing the sum of the scores of these 8 parameters and 5 items by 13. High score indicates low functionality.
Modified Hand Mobility in Scleroderma (mHAMIS) | 3 Months
  It is a method in which the hand functions of individuals are evaluated by a physiotherapist. It evaluates 4 different hand functions based on observation.
Duruoz Hand Index | 3 Months
  Questionnaire form-18 is a likert-type scale that evaluates different hand functions. It can score between 0-90. A high score means a low hand functions.
Six-minute walk test (6MWT) | 3 Months
  In order to evaluate the aerobic capacity of individuals, they will be toured for 6 minutes at a distance of 30 meters. The average 6MWT is between 400 and 700 meters.
Evaluation of muscle strength | 3 Months
  Muscle strength assessment of knee joint flexor and extensor muscle group will be made with Biodex System Pro3® (Biodex Corp, Shirley, NY, USA) device. Before each measurement, patients will be tested 3 times, and knee flexor and extensor maximal concentric isokinetic muscle strength will be measured at 180°/sec 10 repetitions and 60°/sec 5 repetitions angular speeds, with a 30 sec rest interval after each angular velocity.
Evaluation of vascular structure | 3 Months
  Doppler ultrasonography technique is an ultrasonography method that evaluates the blood flow passing through the lumens of the vascular structures in the body. In this method, flow velocity and resistance measurements can be made in vascular structures by measuring the changing return frequencies of sound waves sent from ultrasound probes to the tissues due to the movement of blood cells flowing in the vessel. In the study, the vascular status of the arteries on the forearm and palmar face will be examined by Doppler ultrasonography.
Evaluation of anti-inflammatory effects | 3 Months
  Examination of the cytokine profiles of the patients will be done before and after the treatment for Group 1, and for Group 2 at the initial and final evaluation. IL-6, IL-10, TNF-a and Irisin values, which are the cytokines that the literature focuses on in the pathophysiology of systemic sclerosis, will be checked by blood analysis with the same measurement units at Hacettepe University Central Laboratory.
Hospital Anxiety and Depression Scale (HADS) | 3 Months
  It is a scale that evaluates anxiety and depression, which are psychological symptoms that can occur with diseases, with 14 items. Each question is scored between 0-3 points and a total score between 0 and 21 points can be obtained. A total score of 0-7 is considered normal, a score of 8-10 is considered borderline abnormal (borderline case), and a score of 11-21 is considered abnormal (case).
  0-7 points are normal, 8-10 points are borderline abnormal (borderline case) and 11-21 points are abnormal (case) It is considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)